CLINICAL TRIAL: NCT05219032
Title: Interpreters as Advocates for Hispanic Patients With Hypertension
Brief Title: Interpreters as Advocates for Hypertensive Patients
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Lack of enrollment.
Sponsor: Case Western Reserve University (Other)
Collaborators: National Institute on Minority Health and Health Disparities (NIMHD) (NIH)
Responsible Party: Principal Investigator, Daryl Thornton, Associate Professor, Case Western Reserve University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: P60MD002265DT2; 5P60MD002265-03 (NIH)
Record Dates: First submitted 2021-12-31; First posted 2022-02-01 (Actual); Last update posted 2022-02-01 (Actual); Status verified 2022-01

CONDITIONS: Hypertension
Keywords: Hypertension; Spanish
MeSH Terms: conditions — Hypertension

STUDY DESIGN:
Who Masked: Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Interpreter (Experimental): Professional Spanish interpreter
  Interventions: Behavioral: Professional Medical Interpreter
- Usual Care (No Intervention): Usual care provided to patients

INTERVENTIONS:
Behavioral: Professional Medical Interpreter — A professional medical interpreter accompanies patient to each appointment.
  Arms: Interpreter

SUMMARY:
The purpose of the study is to determine if medical interpreters trained to advocate on behalf of their patients deliver improved care compared to standard medical interpreters

DETAILED DESCRIPTION:
Over 21 million Americans have limited English proficiency. About two-thirds of these individuals speak Spanish. Limited English proficiency has major adverse impacts on health and health care. Using trained medical interpreters may help overcome this language barrier. Compared to patients who need but don't get an interpreter, patients who use trained medical interpreters have better satisfaction, quality of care, and health outcomes. However, the outcomes of patients using interpreters is often poorer than that of English-speaking patients. This randomized controlled trial will test the utility of using interpreters as advocates for Spanish-speaking inner city patients with hypertension.

ELIGIBILITY:
Inclusion Criteria:

* Spanish speaking
* Limited English proficiency
* Uncontrolled hypertension
* Regular visit with primary care provider who is not proficient in Spanish

Exclusion Criteria:

-

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 38 (Actual)
Dates: Start 2010-04 (Actual); Primary Completion 2012-12 (Actual); Study Completion 2014-01 (Actual)

PRIMARY OUTCOMES:
Patient reported satisfaction with the clinical encounter with their clinician | 6 months
  Patients will rate their satisfaction with the clinical encounter with their clinician y responding to several questions about the encounter using a 5-point Likert scale.

SECONDARY OUTCOMES:
Provider reported satisfaction with the clinical encounter with the patient | 6 months
  Providers will rate their satisfaction with the clinical encounter with the patient by responding to several questions about the encounter using a 5-point Likert scale.
Change in systolic and diastolic blood pressure | 6 months
  Net change in systolic and diastolic blood pressure